CLINICAL TRIAL: NCT03844841
Title: DExmEdetomidine Sedation Versus Propofol SEDATION FOR Catheter ABLATION of Atrial Fibrillation Under a Cardiologist Supervision: A Randomized Controlled Pilot STUDY
Brief Title: The Deep Sedation for Ablation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-02128
Record Dates: First submitted 2018-10-30; First posted 2019-02-19 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation; Ablation; Sedation; Propofol; Dexmedetomidine
Keywords: Atrial Fibrillation; Ablation; Sedation; Anesthesia; Propofol; Dexmedetomidine
MeSH Terms: conditions — Atrial Fibrillation | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol (Active Comparator): Active agent: Propofolum (2,6-Diisopropylphenol). Route of administration: intravenous
  Interventions: Drug: Propofol
- Dexmedetomidine (Active Comparator): Active agent: Dexmedetomidinum ut Dexmedetomidini hydrochloridum. Route of administration: intravenous
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — At minimum 5 minutes before start of sedation for atrial fibrillation ablation a bolus of fentanyl (20-50 µg) will be administered. Thereafter, sedation is induced via the continuous infusion of propofol using a target-controlled infusion (TCI) pump. The effect-site propofol concentration will be initially set to 1.5 µg/ml, unless the patient is already sedated by fentanyl. Subsequently, an effect-site propofol concentration of 1 µg/ml will be chosen adjusted stepwise (using steps of 0.3 µg/ml) to reach a target score of 2-3 on the MOAA/S scale. In case of pain fentanyl can be administered bolus-wise (10-30 µg) at the cardiologists discretion.
  Arms: Propofol
Drug: Dexmedetomidine — At minimum 5 minutes before start of sedation for atrial fibrillation ablation a bolus of fentanyl (20-50 µg) will be administered. Thereafter, sedation is induced with a loading dose of dexmedetomidine (0.8 µg/kg) over 10 minutes. The maintenance dexmedetomidine dose is adjusted to the appropriate sedation criteria for CA (0.4 µg/kg/h) and for a target score of 2-3 on the MOAA/S scale. In case of pain, additional fentanyl can be administered bolus-wise (10-30 µg) at the cardiologists discretion.
  Arms: Dexmedetomidine

SUMMARY:
Catheter ablation (CA) is an established therapeutic option for patients with symptomatic atrial fibrillation (AF). During the procedure, patients are usually sedated and analgesized, most commonly by administration of Propofol combined with opioids under the supervision of the electrophysiologist. However, due to the depressive effect of Propofol on the respiratory system, this regimen is not without risk. Dexmedetomidine is a highly selective alpha 2 agonist that demonstrates both analgesic and hypnotic properties with only weak effect on the respiratory system. The pharmacological profile of Dexmedetomidine may be advantageous for sedation during CA of AF. The aim of this randomized trial is to test this hypothesis and explore the safety and efficacy of Dexmedetomidine during CA of AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia. In symptomatic patients, electroanatomic mapping aided catheter ablation (CA) is an established therapeutic option. The intervention may last several hours, during which patients are required to lie as still as possible, as inadequate patient movements disturb the electroanatomic map, prolong the intervention and increase its complication risks. Therefore patients are usually sedated and analgesized, most commonly by administration of Propofol combined with opioids under the supervision of the electrophysiologist. Despite its wide use, this regimen is not without risk, as Propofol has a pronounced depressive effect on the respiratory system.

Dexmedetomidine is a highly selective alpha 2 agonist that demonstrates both analgesic and hypnotic properties with only weak respiratory depression. By reducing sympathetic activity it also reduces the stress response to an intervention. For these reasons, Dexmedetomidine is commonly used in intensive care units, where it has been shown to be well tolerated. Consequently, its range of application has been increasingly widened and good experience has been made with its use in transfemoral valve replacement procedures or gastroenterological interventions.

The pharmacological profile of dexmedetomidine may be also advantageous for sedation during CA of AF. The aim of this randomized trial is to test this hypothesis and explore the safety and efficacy of Dexmedetomidine during CA of AF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Informed consent as documented by signature
* Catheter ablation of atrial fibrillation at the Department of Cardiology, Inselspital Bern

Exclusion Criteria:

* Contraindication to sedation by the electrophysiologist
* Contraindications to either propofol or dexmedetomidine sedation
* Contraindication for targeted controlled propofol infusion (BMI > 35)
* American Society of Anesthesiologists (ASA) classification > III
* Advanced heart block (second or third degree), if no pacemaker or internal cardioverter defibrillator is implanted
* Arterial hypotension (mean < 80 mmHg)
* Severe heart failure (LVEF ≤ 30%)
* Indication for general anaesthesia
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Combined Incidence of Sedation-Emergent Adverse Events (Combined Safety Endpoint) | within 24 hours after completion of procedure
  * Number of participants with sustained bradycardia necessitating cardiac pacing
  * Number of participants with Hypercapnia, defined as rise of transcutaneously measured carbon dioxide levels (tcCO2) > 20mmHg
  * Number of participants with Oxygen desaturation (<90%) necessitating assisted ventilation or further airway management in any form (including chin lift, oropharyngeal airway, bag, and mask ventilation or intubation)
  * Number of participants with Hypotension necessitating termination of sedation or vasopressor administration
  * Number of participants with necessity of termination or change of sedation protocol
  * Number of participants with aborted procedure due to sedation issues

SECONDARY OUTCOMES:
Incidence of Sedation-Emergent Adverse Events (Individual Safety Endpoints) | within 24 hours after completion of procedure
  All single components of the primary endpoint
Other complications | from start until end of ablation procedure
  Number of complications not related to sedation (cardiac tamponade, stroke/transient ischemic attack, pericardial effusion necessitating therapeutic intervention, bleeding necessitating therapeutic intervention, others) [number of events]
Opiod dose | from start until end of ablation procedure
  Opiod dose required for analgesia [ug]
Procedure duration | from start until end of ablation procedure
  Total duration of the procedure [minutes]
Fluoroscopy time | from start until end of ablation procedure
  Duration of fluoroscopy [minutes]
General sedation efficacy: occurrence and number of shiftings | from start until end of ablation procedure
  General sedation efficacy assessed by the occurrence and number of shiftings of the acquired 3D map due to patient movements, necessitating remapping [number of events]
Sedation depth | from start until end of ablation procedure
  Depth of sedation assessed by the Modified Observer's Alertness/Sedation (MOAA/S) scale [mean score]
Blood pressure | from start until end of ablation procedure
  Mean systolic, diastolic and mean blood pressure during sedation and mean drop of blood pressure (pre-procedural blood pressure minus mean blood pressure during sedation) [mmHg]
Heart rate | from start until end of ablation procedure
  Mean heart rate during sedation and mean drop of heart rate (pre-procedural heart rate minus mean heart rate during sedation) [beats per minute]
Refractory period | from start until end of ablation procedure
  Effective refractory period of the atria and atrioventricular node [ms]
Wenckebach point | from start until end of ablation procedure
  Wenckebach point of the atrioventricular node [ms]
Arrhythmia inducibility | from start until end of ablation procedure
  Rate of inducibility of supraventricular arrhythmias during pacing manoeuvres (number of successful/number of attempts) [%]
Patient satisfaction: Patient Satisfaction with Sedation Instrument (PSSI) [score] | within 24 hours after completion of procedure
  Patient satisfaction as assessed by the Patient Satisfaction with Sedation Instrument (PSSI) [score]
Cardiologist satisfaction: Clinician Satisfaction with Sedation Instrument (CSSI) [score] | within 24 hours after completion of procedure
  Cardiologist satisfaction as assessed by the Clinician Satisfaction with Sedation Instrument (CSSI) [score]

CONTACTS AND LOCATIONS:
Overall Officials: Helge Servatius, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Department of Cardiology, University Hospital Inselspital Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Servatius H, Kueffer T, Erdoes G, Seiler J, Tanner H, Noti F, Haeberlin A, Madaffari A, Branca M, Dutschler S, Theiler L, Reichlin T, Roten L. Electrophysiological differences of randomized deep sedation with dexmedetomidine versus propofol. BMC Anesthesiol. 2024 Jul 31;24(1):263. doi: 10.1186/s12871-024-02647-x. PMID 39085782